CLINICAL TRIAL: NCT00143312
Title: Prospective, Open-Label, Non-Comparative, Multicenter Study for the Secondary Prophylaxis of Invasive Fungal Infections (IFI) With Voriconazole in Patients With Allogeneic Stem Cell Transplants (SCT).
Brief Title: Voriconazole for Secondary Prophylaxis of Invasive Fungal Infections in Patients With Allogeneic Stem Cell Transplants
Acronym: VOSIFI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A1501038
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2009-06-01 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-09

CONDITIONS: Prophylaxis Of Invasive Fungal Infections
Keywords: Invasive Fungal Infection, Allogenic Stem Cell Transplant, prophylaxis, leukemia, voriconazole
MeSH Terms: conditions — Invasive Fungal Infections; Leukemia | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: voriconazole

INTERVENTIONS:
Drug: voriconazole — Voriconazole is given to patients at least 48 hours after chemotherapy

SUMMARY:
To prevent recurrence of invasive fungal infection in patients with allogeneic stem cell transplants

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven or probable IFI in previous 12 months receiving an allogenic stem cell transplant for any haematological disease

Exclusion Criteria:

* Pregnant or lactating women
* Severe disease other tham the underlying condition
* Active, symptomatic uncontrolled Invasive Fungal Infection
* Any evidence of active fungal disease as defined by MSG-EORTC criteria
* Concomitant use of Voriconazole 36 hours before chemotherapy until 48 hours after chemotherapy
* Other medical conditions, including HIV positive serology that would interfere with the evaluation of therapeutic response or safety of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Pfizer Investigational Site, Leuven, Belgium
- France (5):
  - Pfizer Investigational Site, Marseille, Cedex 09
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Pessac
  - Pfizer Investigational Site, Strasbourg
- Germany (3):
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Würzburg
- Pfizer Investigational Site, Lisbon, Lisbon District, Portugal
- Spain (2):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
- Pfizer Investigational Site, Stockholm, Sweden
- Pfizer Investigational Site, Ch-4031 Basel, Switzerland
- United Kingdom (2):
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501038&StudyName=Voriconazole%20for%20Secondary%20Prophylaxis%20of%20Invasive%20Fungal%20Infections%20in%20Patients%20with%20Allogeneic%20Stem%20Cell%20Transplants

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects with proven or probable Invasive Fungal Infection (IFI) in the previous 12 months, who were receiving an allogeneic Stem Cell Transplant (SCT) for any hematologic disease, were enrolled into the study if all other inclusion/exclusion criteria were met.
Groups:
- Voriconazole: All subjects received voriconazole as study medication for prophylaxis, for a minimum of 100 days after transplant. Subjects received an intravenous (IV; 6 mg/kg)) or oral (PO; 400 mg) loading dose every 12 hours (q12h) for 2 doses, followed by maintenance (i.e., prophylactic) doses of 4 mg/kg IV q12h or 200 mg PO q12h, if the subject weighed ≥40 kg. If the subject weighed <40 kg, the PO loading dose was 200 mg PO q12h for 2 doses, followed by maintenance doses of 100 mg PO q12h.
Period: Overall Study
Arm/Group | Voriconazole
Started | 45
Completed | 29
Not Completed | 16
Not completed — Death | 11
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Other | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Voriconazole
Number analyzed (Participants) | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 48.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Proven or Probable Invasive Fungal Infection (IFI): Start of Prophylaxis Until 12-month Follow-up Visit
Description: Number of participants developing a proven or probable IFI from start of voriconazole prophylaxis until 12-month follow up
Time Frame: 12 months
Population: Complete case analysis (ie, outcome must be observed and/or subject must be evaluable for entire period of interest) using modified intent-to-treat (MITT) population (ie, subjects had at least 1 dose of voriconazole & at least 1 post-enrollment efficacy assessment & previous diagnosis of proven or probable IFI, confirmed by Data Review Committee).
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 30
participants | 3
Statistical Analysis 1: Comparison: Voriconazole; Test type: Superiority or Other; Crude IFI Rate (percent) at 12 months = 7, 95% CI [2 to 19]
Statistical Analysis 2: Comparison: Voriconazole; Test type: Superiority or Other; IFI Rate (percent) at 12 months = 10, 95% CI [2 to 27]

2. Secondary Outcome: Occurrence of Proven or Probable Invasive Fungal Infection (IFI): Start of Prophylaxis Until 6-month Follow-up Visit
Description: Number of participants developing a proven or probable IFI from start of voriconazole prophylaxis until 6-month follow up
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 34
participants | 3
Statistical Analysis 1: Comparison: Voriconazole; Test type: Superiority or Other; IFI Rate (percent) at 6 months = 8.82, 95% CI [2 to 24] — Exact 95% Confidence Interval For Proportion; Expressed as a percentage

3. Secondary Outcome: Occurrence of Proven or Probable Invasive Fungal Infection (IFI): Start of Voriconazole Prophylaxis Until End of Prophylaxis Visit
Description: Number of participants developing a proven or probable IFI from start of voriconazole prophylaxis until the End of Prophylaxis visit
Time Frame: 150 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 34
participants | 3
Statistical Analysis 1: Comparison: Voriconazole; Test type: Superiority or Other; IFI Rate (percent) at End of Prophylaxis = 8.82, 95% CI [2 to 24] — Exact 95% Confidence Interval For Proportion; Expressed as a percentage

4. Secondary Outcome: Time to Occurrence of Proven or Probable Invasive Fungal Infection (IFI)
Description: Time to occurrence of proven or probable IFI from the start of voriconazole prophylaxis. Time to occurrence is strictly time to recorded diagnosis of IFI since the exact day on which the IFI began will not be known.
Time Frame: 12 months
Population: Modified intent-to-treat (MITT) population (considered evaluable for efficacy) consisted of all subjects who had at least 1 dose of voriconazole & at least 1 post-enrollment efficacy assessment & had a previous diagnosis of proven or probable IFI, confirmed by the Data Review Committee. Three subjects in the MITT population experienced an IFI.
Measure: Number; unit: days
Arm/Group | Voriconazole
Number analyzed (Participants) | 42
days
  time to recurrent IFI (first subject) | 6
  time to recurrent IFI (second subject) | 22
  time to recurrent IFI (third subject) | 81

5. Secondary Outcome: Time to Occurrence of Proven or Probable New (New Pathogen) Invasive Fungal Infection (IFI)
Description: Time to occurrence of proven or probable new (new pathogen) IFI from the start of voriconazole prophylaxis. Time to occurrence is strictly time to recorded diagnosis of IFI.
Time Frame: 12 months
Population: Modified intent-to-treat (MITT) population (considered evaluable for efficacy) consisted of all subjects who had at least 1 dose of voriconazole & at least 1 post-enrollment efficacy assessment & had a previous diagnosis of proven or probable IFI, confirmed by the Data Review Committee. One subject in the MITT population experienced a new IFI.
Measure: Number; unit: days
Arm/Group | Voriconazole
Number analyzed (Participants) | 42
days | 81

6. Secondary Outcome: Time to Occurrence of Proven or Probable Recurrent Invasive Fungal Infection (IFI) (Same Pathogen as Previous Baseline IFI)
Description: Time to occurrence of proven or probable recurrent (same pathogen as baseline) IFI from the start of voriconazole prophylaxis. Time to occurrence is strictly time to recorded diagnosis of IFI. The pathogen identified as the positive culture recorded nearest to, but not after, the proven or probable IFI, was assumed to be responsible for the IFI.
Time Frame: 12 months
Population: Modified intent-to-treat (MITT) population (considered evaluable for efficacy) consisted of all subjects who had at least 1 dose of voriconazole & at least 1 post-enrollment efficacy assessment & had a previous diagnosis of proven or probable IFI, confirmed by the Data Review Committee. Two subjects experienced a recurrent proven or probable IFI.
Measure: Number; unit: days
Arm/Group | Voriconazole
Number analyzed (Participants) | 42
days
  time to IFI (first subject) | 6
  time to IFI (second subject) | 22

7. Secondary Outcome: Survival Without Proven or Probable Invasive Fungal Infection (IFI)
Description: Number of participants who survive (ie., are alive) without proven or probable IFI at each of the 6 and 12 month follow-up visits
Time Frame: 6 months, 12 months
Population: Complete case analysis using MITT population (ie, all subjects who had at least 1 dose of study medication & at least 1 post-enrollment efficacy assessment & a previous diagnosis of proven or probable IFI, confirmed by Data Review Committee) & either provided an IFI assessment at follow-up visit, died or experienced an IFI before that visit.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 39
participants
  survived free of IFI until 6 months | 31
  survived free of IFI until 12 months | 27
Statistical Analysis 1: Comparison: Voriconazole; Test type: Superiority or Other; survive free of IFI (percent): 6 months = 79, 95% CI [64 to 91] — Exact 95% Confidence Interval For Proportion; Expressed as a percentage
Statistical Analysis 2: Comparison: Voriconazole; Test type: Superiority or Other; survive free of IFI (percent): 12 months = 69, 95% CI [52 to 83] — Exact 95% Confidence Interval For Proportion; Expressed as a percentage

ADVERSE EVENTS:
Arm/Group | Voriconazole
Serious Adverse Events (participants affected / at risk) | 23/45
Other Adverse Events (participants affected / at risk) | 42/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole (N=45)
Abdominal pain (Gastrointestinal disorders) | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atrial fibrillation (Cardiac disorders) | 1
Blood creatine increased (Investigations) | 1
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Diarrhoea infectious (Infections and infestations) | 1
Disease progression (General disorders) | 1
Electrocardiogram change (Investigations) | 1
Encephalitis herpes (Infections and infestations) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Eye swelling (Eye disorders) | 1
Facial paresis (Nervous system disorders) | 1
Graft versus host disease (Immune system disorders) | 2
Haemolysis (Blood and lymphatic system disorders) | 1
Hallucination (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Liver function test abnormal (Investigations) | 1
Loss of consciousness (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 2
Sputum culture positive (Investigations) | 1
Tachycardia (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Venoocclusive disease (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole (N=45)
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6
Acute graft versus host disease (Immune system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 4
Anxiety (Psychiatric disorders) | 3
Asthenia (General disorders) | 4
Chills (General disorders) | 5
Cholestasis (Hepatobiliary disorders) | 3
Chronic graft versus host disease (Immune system disorders) | 3
Conjunctivitis (Eye disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Cytomegalovirus infection (Infections and infestations) | 4
Diarrhoea (Gastrointestinal disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 5
Fatigue (General disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Graft versus host disease (Immune system disorders) | 12
Hallucination (Psychiatric disorders) | 3
Headache (Nervous system disorders) | 13
Hepatotoxicity (Hepatobiliary disorders) | 3
Hypertension (Vascular disorders) | 8
Transfusion reaction (Injury, poisoning and procedural complications) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 7
Liver function test abnormal (Investigations) | 4
Mucosal inflammation (General disorders) | 17
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 3
Oedema peripheral (General disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pyrexia (General disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 6
Sinusitis (Infections and infestations) | 3
Sleep disorder (Psychiatric disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Vomiting (Gastrointestinal disorders) | 13
Weight decreased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.